CLINICAL TRIAL: NCT00833690
Title: A Randomized, Double-blind, Placebo-controlled, Dose-ranging Trial of Oral Inosine to Assess Safety and Ability to Elevate Urate in Early Parkinson's Disease
Brief Title: Safety of Urate Elevation in Parkinson's Disease
Acronym: SURE-PD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Parkinson Study Group (Network)
Collaborators: Massachusetts General Hospital (Other); Harvard School of Public Health (HSPH) (Other); University of Rochester (Other); Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Michael Schwarzschild, Principal Investigator, The Parkinson Study Group
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INO-PD-P2-2008
Record Dates: First submitted 2009-01-27; First posted 2009-02-02 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Parkinson disease; PD; inosine; urate; uric acid; cerebrospinal fluid
MeSH Terms: conditions — Parkinson Disease | interventions — Inosine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- [A:] (Placebo Comparator): Placebo to produce no urate elevation
  Interventions: Drug: Placebo
- [B:] (Experimental): Inosine to produce a mild urate elevation
  500 mg of active substance per capsule; 1 to 6 capsules per day (in up to 3 divided doses) for 2 years; dosing titrated to a mildly elevated serum urate range of 6.1 - 7.0 mg/dL
  Interventions: Drug: inosine
- [C.] (Experimental): Inosine to produce a moderate urate elevation
  500 mg of active substance per capsule; 1 to 6 capsules per day (in up to 3 divided doses) for 2 years; dosing titrated to a moderately elevated serum urate range of 7.1 - 8.0 mg/dL
  Interventions: Drug: inosine

INTERVENTIONS:
Drug: Placebo — 500 mg of inactive substance per capsule; 1 to 6 capsules per day (in up to 3 divided doses) for 2 years; dosing adjusted algorithmically to parallel that in the inosine arms
  Arms: [A:]
Drug: inosine — 500 mg of active substance per capsule; 1 to 6 capsules per day (in up to 3 divided doses) for 2 years; dosing titrated to a mildly elevated serum urate range of 6.1 - 7.0 mg/dL
  Other Names: hypoxanthine 9-β-D-ribofuranoside
  Arms: [B:]
Drug: inosine — 500 mg of active substance per capsule; 1 to 6 capsules per day (in up to 3 divided doses) for 2 years; dosing titrated to a moderately elevated serum urate range of 7.1 - 8.0 mg/dL
  Other Names: hypoxanthine 9-β-D-ribofuranoside
  Arms: [C.]

SUMMARY:
The purpose of this study is to determine the safety and tolerability of inosine and its ability to raise urate levels in blood and cerebral spinal fluid in individuals with early Parkinson disease. This will determine whether it is appropriate to proceed with a larger study of inosine's ability to modify the rate of disability progression in PD.

DETAILED DESCRIPTION:
Background & Rationale:

Convergent epidemiological and clinical observations have identified urate - a major antioxidant and the end product of purine metabolism in humans - as the first molecular predictor of both the risk and the progression of typical Parkinson's disease (PD). Among some 1600 early PD patients enrolled in prior clinical trials, those with baseline serum urate levels in the highest quintile (i.e., in the upper normal range) displayed a 40% slower rate of clinical (disability) progression compared to those with baseline urate at or below the median (with p<0.000001 for trend across quintiles). Similarly, amongst those who underwent serial SPECT brain scans for changes in dopamine transporter (DAT) binding, those with higher baseline serum urate levels displayed a slower rate of radiographic progression (loss of striatal DAT). Moreover, urate levels in baseline cerebrospinal fluid (CSF) samples also correlate inversely with rates of clinical progression. Although this link between urate and a slower decline in PD appears reproducible and robust, the critical question of causality remains to be answered by a well-designed clinical trial. The biological plausibility of neuroprotection by urate strengthens the rationale for expedient pursuit of a trial. The availability of established pharmacological approaches to elevating urate makes such a trial feasible. In particular, inosine, an orally bioavailable, central nervous system (CNS)-penetrant purine precursor of urate, offers a practical strategy as it can readily elevate serum urate, has been widely consumed as a nutritional supplement, and has been administered chronically in several multi-year clinical trials for multiple sclerosis. Before embarking on a neuroprotection trial of inosine for PD, careful assessment of the safety, validity and methodology of this approach in PD patients is warranted.

Specific Aims:

The main goal of the study is to determine whether inosine is suitable for phase III evaluation of its ability to modify the rate of disability progression in PD. Specific primary aims entail the determination of the safety and tolerability of oral inosine, and its ability to elevate urate levels in serum or CSF; and the selection of an optimal dosing regimen. Secondary aims entail the further optimization of a possible phase III study design.

Methods:

A placebo-controlled double-blind dose-ranging randomized trial of inosine will be conducted in early PD. Ninety untreated subjects diagnosed with idiopathic PD and with a serum urate below the population mean (~6 mg/dL) will be enrolled at 17 North American sites and randomized to one of three treatment groups (n=30): 1) placebo, 2) inosine dosed to produce a mild elevation in serum urate, and 3) inosine dosed to produce a moderate elevation. Tolerability, validity (urate elevation), dosage and symptomatic efficacy will be assessed after 12 weeks of treatment. Contingent on adequate tolerability and validity as assessed in this short-term analysis, the study will continue for 2 years total duration with 2 groups (placebo and a merged single inosine dosing group) or the original 3 to assess long-term tolerability and safety, which will focus on main known risks of urolithiasis and gouty arthritis and the theoretical risk of cardiovascular disease.

Significance:

This study will determine whether a phase III trial of inosine as a potential neuroprotectant in PD is warranted. If it is, then the present study could shorten substantially the lead time, and through optimization of key design features would enhance the likelihood of its safety and success.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD with at least two of the cardinal signs of PD (resting tremor, bradykinesia, rigidity)
* Currently not taking or needing any treatment for PD other than an monoamine oxidase-B (MAO-B) inhibitor
* Age 30 or older at the time of PD diagnosis
* Diagnosis of PD made within past 3 years
* Serum urate ≤ 5.8 mg/dL at initial screening

Exclusion Criteria:

* History of kidney stones, gout, stroke, or heart attack
* History of renal disease or certain cardiovascular problems within the past year
* Acidic urine (pH ≤ 5.0), uric acid, or urate crystalluria at screening
* Use of certain medications including co-enzyme Q, creatine, more than 50 IU of vitamin E daily, and more than 300 mg of vitamin C daily. (A standard daily multivitamin is permitted.)
* Use of anti-PD and other medications targeting central nervous system dopamine transmission
* Known unstable medical or psychiatric condition that may compromise participation in the study
* Women who are pregnant or lactating

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Schwarzschild, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (16):
- United States (16):
  - University of Southern California, Los Angeles, California
  - Eastern Connecticut Neurology Specialists, LLC, Manchester, Connecticut
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - Struthers Parkinson's Center, Golden Valley, Minnesota
  - Duke University School of Medicine, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Butler Hospital Movement Disorder Program, Providence, Rhode Island
  - Scott & White Hospital, Temple, Texas

REFERENCES:
- [Derived] Schwarzschild MA, Macklin EA, Bakshi R, Battacharyya S, Logan R, Espay AJ, Hung AY, Bwala G, Goetz CG, Russell DS, Goudreau JL, Parashos SA, Saint-Hilaire MH, Rudolph A, Hare JM, Curhan GC, Ascherio A; Parkinson Study Group SURE-PD Investigators. Sex differences by design and outcome in the Safety of Urate Elevation in PD (SURE-PD) trial. Neurology. 2019 Oct 1;93(14):e1328-e1338. doi: 10.1212/WNL.0000000000008194. Epub 2019 Sep 4. PMID 31484712
- [Derived] Parkinson Study Group SURE-PD Investigators; Schwarzschild MA, Ascherio A, Beal MF, Cudkowicz ME, Curhan GC, Hare JM, Hooper DC, Kieburtz KD, Macklin EA, Oakes D, Rudolph A, Shoulson I, Tennis MK, Espay AJ, Gartner M, Hung A, Bwala G, Lenehan R, Encarnacion E, Ainslie M, Castillo R, Togasaki D, Barles G, Friedman JH, Niles L, Carter JH, Murray M, Goetz CG, Jaglin J, Ahmed A, Russell DS, Cotto C, Goudreau JL, Russell D, Parashos SA, Ede P, Saint-Hilaire MH, Thomas CA, James R, Stacy MA, Johnson J, Gauger L, Antonelle de Marcaida J, Thurlow S, Isaacson SH, Carvajal L, Rao J, Cook M, Hope-Porche C, McClurg L, Grasso DL, Logan R, Orme C, Ross T, Brocht AF, Constantinescu R, Sharma S, Venuto C, Weber J, Eaton K. Inosine to increase serum and cerebrospinal fluid urate in Parkinson disease: a randomized clinical trial. JAMA Neurol. 2014 Feb;71(2):141-50. doi: 10.1001/jamaneurol.2013.5528. PMID 24366103
- See also: Related Info — http://www.Parkinson-Study-Group.org

RESULTS

PARTICIPANT FLOW:
Groups:
- [A:]Placebo: Placebo to produce no urate elevation
- [B:]Mild: Inosine to produce a mild urate elevation
- [C.]Moderate: Inosine to produce a moderate urate elevation
Period: Overall Study
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Started | 25 | 24 | 26
Completed | 21 | 22 | 26
Not Completed | 4 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Discontinued study drug | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate | Total
Number analyzed (Participants) | 25 | 24 | 26 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (11) | 62 (10) | 62 (11) | 62 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 14 | 41
  Male | 12 | 10 | 12 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 25 | 22 | 26 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 0
  White | 24 | 22 | 24 | 70
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 26 | 75
Years since symptom onset [Mean (Standard Deviation); unit: Years] | 2.4 (1.3) | 2.8 (1.9) | 2.2 (2.0) | 2.4 (1.8)
Years since diagnosis [Mean (Standard Deviation); unit: Years] | 1.1 (1.3) | 1.3 (1.0) | 0.6 (0.7) | 1.0 (1.1)
Serum Urate [Mean (Standard Deviation); unit: mg/dL] | 4.5 (0.7) | 4.3 (1.2) | 4.6 (0.9) | 4.5 (0.9)
Serum urate in women [Mean (Standard Deviation); unit: mg/dL] | 4.4 (0.8) | 3.9 (1.3) | 4.4 (0.8) | 4.2 (1.0)
Serum urate in men [Mean (Standard Deviation); unit: mg/dL] | 4.7 (0.5) | 5.0 (0.8) | 4.9 (0.9) | 4.8 (0.7)
United Parkinson's Disease Rating Scale (UPDRS) score total [Mean (Standard Deviation); unit: points] — The UPDRS is designed to monitor disability and impairment due to Parkinson's disease. It comprises several parts. Part I evaluates "Mentation, Behavior, and Mood" (with a maximum of 16 points; more points are worse); Part II evaluates "Activities of Daily Living" (with a maximum of 52 points); Part III entails a "Motor Examination" (with a maximum of 108 points). Total score of Parts I-III sums the points from all parts and thus can range from a minimum of 0 (best) to a maximum of 176 (worst).
  points | 23 (10) | 20 (9) | 21 (10) | 22 (10)
Montreal Cognitive Assessment (MoCA) [Mean (Standard Deviation); unit: Score] — The MoCA assesses short term and working memory, visual-spatial abilities, executive function, attention, concentration, language and orientation. The total score ranges from 0 to 30 (highest function).
  Score | 28 (1.9) | 28 (1.8) | 28 (2.0) | 28 (1.9)
Geriatric Depression Scale-short form (GDS-S) [Mean (Standard Deviation); unit: Score] — GDS-S is a short 15 'yes/no' question instrument for assessing depression in older adults. Questions are answered by the research participant (i.e., self-rater). Scores range range from 0 to 15 and higher scores represent greater depression. Scores of 5-9 and >9 have been correlated with mild and moderate-severe depression, respectively.
  Score | 1.5 (1.9) | 1.4 (1.7) | 1.8 (2.6) | 1.5 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Tolerability
Description: Defined as the extent to which assigned treatment could continue without prolonged dose reduction (>48 consecutive days or >73 cumulative days, which is 10% of total 2-year follow-up) due to adverse experiences (AEs), and was assessed after 6 and 24 months on study drug. Units of measure are percentage points (i.e., % of participants in the group).
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 25 | 24 | 26
percentage of participants | 96 | 96 | 100

2. Primary Outcome: Tolerability
Description: Defined as the extent to which assigned treatment could continue without prolonged dose reduction (>48 consecutive days or >73 cumulative days, which is 10% of total 2-year follow-up) due to AEs, and was assessed after 6 and 24 months on study drug. Units of measure are percentage points (i.e., % of participants in the group).
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 25 | 24 | 26
percentage of participants | 86 | 92 | 96

3. Secondary Outcome: CSF Urate (All Patients)
Description: Urate concentration in cerebrospinal fluid (CSF)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 11 | 15 | 18
mcg/dL | 427 (190) | 544 (148) | 594 (175)

4. Secondary Outcome: CSF Urate (Females)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 5 | 9 | 10
mcg/dL | 285 (69) | 517 (169) | 575 (176)

5. Secondary Outcome: CSF Urate (Males)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 6 | 6 | 8
mcg/dL | 546 (178) | 586 (113) | 619 (184)

6. Secondary Outcome: CSF Urate as a Proportion of Baseline Serum Urate (All Patients)
Description: Although CSF urate was not measured at baseline, the change of CSF urate from baseline may be indirectly estimated by the ratio of CSF urate (at the 12 week visit when a lumbar puncture was performed) to the serum urate measured in the same subject at baseline. Baseline serum urate and CSF urate concentrations are directly correlated with one another (i.e., individuals with higher serum urate concentrations tend to have higher CSF urate concentrations) even though the concentration of urate in CSF is typically ~10% of that in serum. The ratio of CSF urate to baseline serum urate can be expressed as the percentage of the value of urate concentration measured in serum at baseline that is measured in CSF (at week 12).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of baseline serum urate
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 11 | 15 | 18
percentage of baseline serum urate | 9.6 (4.0) | 13.1 (4.0) | 13.4 (4.3)

7. Secondary Outcome: CSF Urate as a Proportion of Baseline Serum Urate (Females)
Description: as for outcome 6
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of baseline serum urate
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 5 | 9 | 10
percentage of baseline serum urate | 6.7 (1.8) | 13.5 (5.0) | 13.3 (5.0)

8. Secondary Outcome: CSF Urate as a Proportion of Baseline Serum Urate (Males)
Description: as for outcome 6
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of baseline serum urate
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 6 | 6 | 8
percentage of baseline serum urate | 12.0 (3.8) | 12.4 (2.2) | 13.4 (3.5)

9. Secondary Outcome: Serum Urate
Description: From blood sample drawn prior to enrollment
Time Frame: Screening Visits, up to 45 days prior to Baseline Visit. Specifically, Screening Visit 1 occurred between day -45 and -4; Screening Visit 2 occurred between day -43 and -2.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 25 | 24 | 26
mg/dL
  Screening Visit 1 | 4.63 (0.62) | 4.28 (0.86) | 4.39 (0.78)
  Screening Visit 2 | 4.78 (0.6) | 4.4 (0.88) | 4.48 (0.75)

10. Secondary Outcome: Serum Urate
Description: From blood sample drawn prior to enrollment
Time Frame: Baseline Visit
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 25 | 23 | 26
mg/dL | 4.54 (0.69) | 4.32 (1.2) | 4.62 (0.86)

11. Primary Outcome: Safety
Description: Defined as absence of serious adverse experiences (SAEs) that warranted terminating an inosine treatment arm or the trial, as determined by the Data and Safety Monitoring Committee.
Time Frame: 24 months
Measure: Number; unit: Events
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 25 | 24 | 26
Events | 11 | 2 | 4

12. Secondary Outcome: Serum Urate
Description: From blood sample drawn after taking study drug that day
Time Frame: Visit 01 (Week 2; 14 +/- 3 days after Baseline Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 25 | 24 | 26
mg/dL | 4.8 (0.65) | 6.44 (1.29) | 6.93 (1.42)

13. Secondary Outcome: Serum Urate
Description: From blood sample drawn after taking study drug that day
Time Frame: Visit 02 (Week 4; 28 +/- 3 days after Baseline Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 24 | 24 | 26
mg/dL | 4.73 (0.65) | 6.58 (0.87) | 7.9 (1.29)

14. Secondary Outcome: Serum Urate
Description: From blood sample drawn after taking study drug that day
Time Frame: Visit 03 (Week 6; 42 +/- 3 days after Baseline Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 24 | 24 | 26
mg/dL | 4.85 (0.77) | 6.69 (0.78) | 7.51 (1.24)

15. Secondary Outcome: Serum Urate
Description: From blood sample drawn after taking study drug that day
Time Frame: Visit 04 (Week 9; 63 +/- 5 days after Baseline Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 24 | 24 | 26
mg/dL | 4.62 (0.58) | 6.81 (1.22) | 7.62 (1.02)

16. Secondary Outcome: Serum Urate
Description: From blood sample drawn before taking study drug that day
Time Frame: Visit 05 (Week 12; 84 +/- 7 days after Baseline Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 24 | 24 | 26
mg/dL | 4.74 (0.59) | 5.85 (1.02) | 6.91 (1.09)

17. Secondary Outcome: Serum Urate
Description: From blood sample drawn after taking study drug that day
Time Frame: Visit 06 (Month 6; 180 +/- 7 days after Baseline Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 24 | 23 | 26
mg/dL | 4.85 (1) | 6.94 (1.6) | 8.27 (0.74)

18. Secondary Outcome: Serum Urate
Description: From blood sample drawn after taking study drug that day
Time Frame: Visit 07 (Month 9; 270 +/- 7 days after Baseline Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 24 | 24 | 26
mg/dL | 4.77 (0.89) | 6.77 (1.51) | 8.06 (1.2)

19. Secondary Outcome: Serum Urate
Description: From blood sample drawn after taking study drug that day
Time Frame: Visit 08 (Month 12; 360 +/- 7 days after Baseline Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 22 | 23 | 24
mg/dL | 4.79 (0.89) | 6.87 (1.05) | 7.41 (0.96)

20. Secondary Outcome: Serum Urate
Description: From blood sample drawn after taking study drug that day
Time Frame: Visit 09 (Month 15; 450 +/- 7 days after Baseline Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 18 | 19 | 22
mg/dL | 4.62 (0.69) | 7.26 (0.96) | 7.64 (1.2)

21. Secondary Outcome: Serum Urate
Description: From blood sample drawn after taking study drug that day
Time Frame: Visit 10 (Month 18; 540 +/- 7 days after Baseline Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 16 | 16 | 17
mg/dL | 4.58 (0.76) | 7 (0.97) | 7.64 (0.98)

22. Secondary Outcome: Serum Urate
Description: From blood sample drawn after taking study drug that day
Time Frame: Visit 11 (Month 21; 630 +/- 7 days after Baseline Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 7 | 11 | 14
mg/dL | 4.6 (0.47) | 7.12 (1.21) | 7.56 (1.08)

23. Secondary Outcome: Serum Urate
Description: From blood sample drawn after taking study drug that day
Time Frame: Visit 12 (Month 24; 720 +/- 7 days after Baseline Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 5 | 10 | 9
mg/dL | 4.41 (0.99) | 6.84 (0.76) | 7.19 (1.19)

24. Secondary Outcome: Serum Urate
Description: From blood sample drawn after taking study drug that day
Time Frame: End of Study Drug Visit (ESD) (Month 9-24; 263-727 days after Baseline Visit)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 24 | 24 | 26
mg/dL | 4.66 (0.79) | 6.48 (1.25) | 7.55 (1.6)

25. Secondary Outcome: Serum Urate
Description: From blood sample drawn a month after stopping study drug
Time Frame: Safety Visit (SV); 30 +/- 3 days following ESD or Month 24 Visit
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 24 | 23 | 26
mg/dL | 4.74 (0.77) | 4.69 (1.28) | 4.38 (0.78)

26. Secondary Outcome: Change in Serum Urate
Description: Change from an Average of Baseline and Screening Visits
Time Frame: Visit 01 from Baseline (i.e., between -45 days and +2 weeks)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 25 | 24 | 26
mg/dL | 0.15 (0.41) | 2.1 (0.83) | 2.44 (1.07)

27. Secondary Outcome: Change in Serum Urate
Description: Change from an Average of Baseline and Screening Visits
Time Frame: Visit 02 from Baseline (i.e., between -45 days and +4 weeks)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 24 | 24 | 26
mg/dL | 0.09 (0.48) | 2.24 (1.13) | 3.41 (1.22)

28. Secondary Outcome: Change in Serum Urate
Description: Change from an Average of Baseline and Screening Visits
Time Frame: Visit 03 from Baseline (i.e., between -45 days and +6 weeks)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 24 | 24 | 26
mg/dL | 0.22 (0.51) | 2.35 (1.03) | 3.02 (1.13)

29. Secondary Outcome: Change in Serum Urate
Description: Change from an Average of Baseline and Screening Visits
Time Frame: Visit 04 from Baseline (i.e., between -45 days and +9 weeks)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 24 | 24 | 26
mg/dL | -0.02 (0.35) | 2.47 (1.34) | 3.13 (1.16)

30. Secondary Outcome: Change in Serum Urate
Description: Change from an Average of Baseline and Screening Visits
Time Frame: Visit 05 from Baseline (i.e., between -45 days and +12 weeks)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 24 | 24 | 26
mg/dL | 0.1 (0.42) | 1.51 (0.8) | 2.42 (1.08)

31. Secondary Outcome: Change in Serum Urate
Description: Change from an Average of Baseline and Screening Visits
Time Frame: Visit 06 from Baseline (i.e., between -45 days and +6 months)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 24 | 23 | 26
mg/dL | 0.21 (0.86) | 2.55 (1.4) | 3.78 (0.95)

32. Secondary Outcome: Change in Serum Urate
Description: Change from an Average of Baseline and Screening Visits
Time Frame: Visit 07 from Baseline (i.e., between -45 days and +9 months)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 24 | 24 | 26
mg/dL | 0.14 (0.68) | 2.43 (1.56) | 3.56 (1.51)

33. Secondary Outcome: Change in Serum Urate
Description: Change from an Average of Baseline and Screening Visits
Time Frame: Visit 08 from Baseline (i.e., between -45 days and +12 months)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 22 | 23 | 24
mg/dL | 0.2 (0.78) | 2.46 (1.24) | 2.96 (1.28)

34. Secondary Outcome: Change in Serum Urate
Description: Change from an Average of Baseline and Screening Visits
Time Frame: Visit 09 from Baseline (i.e., between -45 days and +15 months)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 18 | 19 | 22
mg/dL | 0 (0.67) | 2.9 (0.98) | 3.19 (1.18)

35. Secondary Outcome: Change in Serum Urate
Description: Change from an Average of Baseline and Screening Visits
Time Frame: Visit 10 from Baseline (i.e., between -45 days and +18 months)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 16 | 16 | 17
mg/dL | -0.07 (0.43) | 2.49 (1.07) | 3.26 (1.25)

36. Secondary Outcome: Change in Serum Urate
Description: Change from an Average of Baseline and Screening Visits
Time Frame: Visit 11 from Baseline (i.e., between -45 days and +21 months)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 7 | 11 | 14
mg/dL | -0.07 (0.59) | 2.53 (1.12) | 3.11 (1.46)

37. Secondary Outcome: Change in Serum Urate
Description: Change from an Average of Baseline and Screening Visits
Time Frame: Visit 12 from Baseline (i.e., between -45 days and +24 months)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 5 | 10 | 9
mg/dL | -0.29 (1.08) | 2.22 (0.96) | 2.93 (1.38)

38. Secondary Outcome: Change in Serum Urate
Description: Change from an Average of Baseline and Screening Visits
Time Frame: Safety Visit (SV) from Baseline (i.e., between -45 days and +760 days [+1 month after ESD Visit])
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 24 | 23 | 26
mg/dL | 0.1 (0.62) | 0.35 (0.88) | -0.11 (0.61)

39. Secondary Outcome: Change in Serum Urate
Description: Change from Last Visit on Study Drug
Time Frame: Safety Visit (SV) from End of Study Drug Visit (ESD); i.e., between +263 and +760 days)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Number analyzed (Participants) | 23 | 23 | 26
mg/dL | 0.12 (0.51) | -1.8 (1.33) | -3.2 (1.63)

ADVERSE EVENTS:
Arm/Group | [A:]Placebo | [B:]Mild | [C.]Moderate
Serious Adverse Events (participants affected / at risk) | 9/25 | 2/24 | 4/26
Other Adverse Events (participants affected / at risk) | 18/25 | 22/24 | 20/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [A:]Placebo (N=25) | [B:]Mild (N=24) | [C.]Moderate (N=26)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Human ehrlichiosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [A:]Placebo (N=25) | [B:]Mild (N=24) | [C.]Moderate (N=26)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (4) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2) | 4 (6)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 1 (1) | 3 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 2 (3) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory track infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No